CLINICAL TRIAL: NCT05045794
Title: A Multicenter, Prospective, Open-label, Randomized Controlled Clinical Trial to Compare the Safety and Effectiveness of the VitaSmart Liver Machine Perfusion System With Static Cold Storage for Organ Preservation Prior to Liver Transplantation
Brief Title: Bridge to HOPE: Hypothermic Oxygenated Perfusion Versus Cold Storage Prior to Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bridge to Life Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-2020-01vs
Record Dates: First submitted 2021-08-31; First posted 2021-09-16 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: End Stage Liver DIsease; Liver Failure
Keywords: Hypothermic oxygenated machine perfusion; Liver preservation; Liver transplantation
MeSH Terms: conditions — End Stage Liver Disease; Liver Failure

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label, sequential assignment, non-inferiority design comparing two treatment arms (HOPE, static cold storage)
Masking Description: A centralized radiologist who evaluates imaging (MRCP) for one of the secondary endpoints (ischemic cholangiopathy) will be blinded to treatment assignment. The study is otherwise open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hypothermic oxygenated perfusion (HOPE) (Experimental): Ex-vivo donor liver preservation using static cold storage followed by HOPE using the VitaSmart Liver Machine
  Interventions: Device: VitaSmart Liver Machine Perfusion System; Other: Static cold storage
- Static cold storage (Other): Ex-vivo donor liver preservation using static cold storage only
  Interventions: Other: Static cold storage

INTERVENTIONS:
Device: VitaSmart Liver Machine Perfusion System — Following donor liver retrieval, preservation using static cold storage, and back table preparation in the transplant center operating room, the organ will be flushed with Belzer UW Machine Perfusion Solution (MPS) and perfused through the cannulated portal vein using cold, actively oxygenated MPS that is circulated at low pressure for 90 minutes to 5 hours. After disconnection from the device, donor liver implantation and reperfusion will proceed in accordance with institutional care standards.
  Other Names: VitaSmart Liver Machine; Hypothermic oxygenated perfusion
  Arms: Hypothermic oxygenated perfusion (HOPE)
Other: Static cold storage — Donor liver retrieval and preservation using standard of care cold storage methods

SUMMARY:
This is a prospective, multi-center, controlled, randomized, pivotal study to evaluate the safety and effectiveness of the VitaSmart Liver Machine Perfusion System by comparing clinical outcomes in patients undergoing liver transplantation with ex-vivo liver preservation using static cold storage (SCS) followed by hypothermic oxygenated machine perfusion (HOPE) versus SCS only.

DETAILED DESCRIPTION:
Patients on the UNOS waiting list for liver transplantation who have been consented, meet study eligibility criteria and are matched to a liver allograft from donation after brain death (DBD) or donation after circulatory death (DCD) that meet the extended risk eligibility criteria will be randomized 1:1 to SCS followed by HOPE (HOPE arm) or to SCS only (SCS arm). The objective of the study is to demonstrate the safety and effectiveness of the VitaSmart Liver Machine by comparing endpoints between the HOPE and SCS arms.

Following transplantation, patients will be monitored daily (labs, adverse events, medications/procedures) while inpatient, and then additionally on Days 14 and 30 and Months 3, 6 and 12. The primary efficacy endpoint of early allograft dysfunction (EAD) rate will be assessed between HOPE and control using a non-inferiority design. An interim analysis is planned after approximately 70% of patients have been completed primary endpoint data collection to assess for early study completion based on non-inferiority or superiority.

ELIGIBILITY:
Donation after Brain Death (DBD) Liver Inclusion Criteria (one or more):

* Donor age 50-85 years
* Anticipated cold ischemia time 10-15 hours (excluding HOPE duration)
* Macrosteatosis 10-40%
* Terminal ALT 250-1500 IU/ml
* Peak ALT within 3 days 1000-3000 IU/ml
* Terminal total bilirubin 2-4 mg/dl

Donation after Brain Death (DBD) Liver Exclusion Criteria (one or more):

* Donor age <18 or >85 years
* Anticipated cold ischemia >15 hours
* Macrosteatosis >40%
* Terminal ALT >1500 IU/ml
* Peak ALT within 3 days >3000 IU/ml
* Terminal total bilirubin >4 mg/dl
* Presence of hemodynamic and/or anatomical donor abnormalities that, in the opinion of the Investigator, make the liver allograft unsuitable for transplant into the recipient subject
* Liver intended for split transplant
* Liver from living donor
* Donor terminal serum Na >160 mmol/L

Donation after Cardio-circulatory Death (DCD) Liver Inclusion Criteria (all):

* Donor age 18-60 years
* Anticipated cold ischemia time <12 hours (excluding HOPE duration)
* Functional warm ischemia time ≤35 minutes, defined as interval from the time of onset of donor hypotension (MAP <50mmHg) until the time of donor cross clamp
* Macrosteatosis ≤20%
* Terminal ALT ≤500 IU/ml
* Peak ALT within 3 days ≤2000 IU/ml
* Terminal total bilirubin ≤3 mg/dl

Donation after Cardio-circulatory Death (DCD) Liver Exclusion Criteria (one or more):

* Presence of hemodynamic and/or anatomical donor abnormalities that, in the opinion of the Investigator, make the liver allograft unsuitable for transplant into the recipient subject
* Liver intended for split transplant
* Liver from living donor
* Donor terminal serum Na >160 mmol/L

Recipient Inclusion Criteria (one or more):

* Subject (or legally authorized representative) is able to provide informed consent and HIPAA authorization
* Subject is male or female and at least 18 years of age
* Subject is registered as an active liver recipient on the UNOS waiting list for liver transplantation
* Subject will undergo primary liver transplantation
* Subject is willing to comply with the study requirements and procedures
* Subject with hepatocellular carcinoma as indication for Orthotopic Liver Transplantation; the tumor must be within Milan Criteria or down-staged to Milan Criteria

Recipient Exclusion Criteria (one or more):

* Subject will undergo multiple organ transplantations (liver-kidney, liver-lung, etc.)
* Subject is listed for liver transplantation due to fulminant liver failure (UNOS status 1A)
* Subject is pregnant
* Subject is on respiratory (ventilator dependent) and/or cardiocirculatory support (requires at least one intravenous inotrope to maintain hemodynamics)
* Subject is enrolled in an interventional clinical trial with an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with early allograft dysfunction (EAD) | At Day 7 post-transplant

SECONDARY OUTCOMES:
Model for early allograft function (MEAF) score | Within 3 days post-transplant
  Based on definition by Olthoff et al, 2010 (doi: 10.1002/lt.22091)
Proportion of patients with primary non-function (PNF) | Within 7 days post-transplant
  Based on definition by Pareja et al, 2015 (doi: 10.1002/lt.23990)
Length of hospital stay | Up to study participation ends at 1-year follow-up
  Duration from initial ICU admission to hospital discharge order (measured in days)
Length of intensive care unit stay | Up to study participation ends at 1-year follow-up
  Duration from initial ICU admission to ICU discharge order (measured in days)
Duration on dialysis | Up to study participation ends at 1-year follow-up
  Duration from establishment of graft reperfusion until discontinuation of dialysis (measured in days)
Donor liver utilization rate | Up to study participation ends at 1-year follow-up
Patient survival rate | 30 days, 6 months, 1 year post-transplant
Graft survival rate | 30 days, 6 months, 1 year post-transplant
Incidence of adverse events (AEs) | 1 year post-transplant
Incidence of serious AEs (SAEs) | 1 year post-transplant
Incidence of unanticipated adverse device effects (UADEs) | 1 year post-transplant
Incidence of ischemic cholangiopathy | 6 months, 1 year post-transplant
Incidence of biopsy-proven liver rejection | 6 months, 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: David Reich, MD, Principal Investigator — Drexel University
Locations (16):
- United States (16):
  - Loma Linda University Medical Center, San Bernardino, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Cleveland Clinic, Weston, Florida
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University St. Louis, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SC, Foley DP. Strategies to Improve the Utilization and Function of DCD Livers. Transplantation. 2024 Mar 1;108(3):625-633. doi: 10.1097/TP.0000000000004739. Epub 2023 Jul 27. PMID 37496117